CLINICAL TRIAL: NCT03055637
Title: Evaluation of the Incidence of Palatal Fistula in Furlow Double-opposing Z-plasty vs. Two-flap Palatoplasty for Cleft Palate Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sarah Moustafa Mahmoud Fahmy El-Youtti (Other)
Responsible Party: Sponsor-Investigator, Sarah Moustafa Mahmoud Fahmy El-Youtti, Sarah moustafa mahmoud fahmy Al-Ayoutti, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 28902051202049
Record Dates: First submitted 2017-02-14; First posted 2017-02-16 (Actual); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Fistula of Soft Palate (Disorder)

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with isolated cleft palate (Active Comparator): Patients requiring isolated cleft palate repair
  Interventions: Procedure: Furlow double opposing z-plasty; Procedure: Two flap palatoplasty
- Patients with isolated cleft palate (Active Comparator): Patients requiring isolated cleft palate repair
  Interventions: Procedure: Furlow double opposing z-plasty; Procedure: Two flap palatoplasty

INTERVENTIONS:
Procedure: Furlow double opposing z-plasty — * Furlow, (1986) has described a technique for palatoplasty combining the principles of mucosal lengthening with creation of an intact muscular sling in the palate with double opposing Z-plasty. On the soft palate, mirror image Z-plasties are drawn, one for the nasal musoca and the other oral flaps, the nasal flaps are developed and closed first .The oral flaps are then approximated. The defect created usually closes readily. The closure lines of the two soft plate layers do not overlap, minimizing the potential for contracture. Also, this repair permits closure of the hard palate without lateral incisions
Procedure: Two flap palatoplasty — design the 2-flap palatoplasty, with a 2-layer closure in the hard palate and 3-layer closure in the soft palate,

SUMMARY:
Evaluation of the incidence of palatal fistula in Furlow double-opposing z-plasty versus two-flap palatoplasty for cleft palate repair.

DETAILED DESCRIPTION:
Up to 6 hours before the scheduled arrival time, formula-fed babies may be given formula. Up to 4 hours before the scheduled arrival time, breastfed babies may nurse. Up to 2 hours before the scheduled arrival time, give only clear liquids. Clear liquids include water, Pedialyte®, Kool-Aid® and juices you can see through, such as apple or white grape juice. In the 2 hours before the scheduled arrival time, give nothing to eat or drink. Induction of general anaesthesia will be administered followed by local anaethesia. Then, Surgical prodecure will be done either following the conventional two flap palatoplasty technique or the Furlow double-opposing z-plasty technique.

ELIGIBILITY:
Inclusion Criteria:

1. Age of Repair from 9 to 12 months.
2. Isolated Cleft Palate
3. Operation time should nearly be the same for all patients
4. Surgical skills done by same surgeon
5. Both sexes

Exclusion Criteria:

1. Patients with hypoplasia of palatal tissue.
2. Patients with associated anomalies.
3. Patients with associated syndromes.
4. Other types of cleft palate.

Ages: 9 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2017-02-19 (Estimated); Primary Completion 2017-05-19 (Estimated); Study Completion 2017-05-19 (Estimated)

PRIMARY OUTCOMES:
Incidence of fistula | 6 months